CLINICAL TRIAL: NCT05473585
Title: Impact of New Standards for Tobacco Products Among Dual E-Cigarette/Combusted Cigarette Users - Project 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro00105539; 5R01DA048454 (NIH)
Record Dates: First submitted 2022-07-13; First posted 2022-07-26 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Smoking; Smoking, Cigarette; E-Cig Use; Nicotine Dependence
Keywords: Nicotine Reduction; Dual users
MeSH Terms: conditions — Smoking; Cigarette Smoking; Vaping; Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Participants will complete 4 experimental sessions. At each session, they will receive a different combination of e-cigarette and combusted cigarette.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Study EC + UB CC (Active Comparator): Participants will make choices between the study e-cigarette (EC) device with tobacco flavor and their usual brand (UB) combusted cigarette (CC)
  Interventions: Other: Study e-cigarette
- Study EC + NNC CC (Active Comparator): Participants will make choices between the study EC device with tobacco flavor and the normal nicotine content (NNC) investigational CC
  Interventions: Other: normal nicotine content cigarettes; Other: Study e-cigarette
- Study EC + VLNC CC (Experimental): Participants will make choices between the study EC device with tobacco flavor and the very low nicotine content (VLNC) investigational CC
  Interventions: Other: very low nicotine content cigarettes; Other: Study e-cigarette
- Own EC + UB CC (No Intervention): Participants will make choices between their own EC device with their own tobacco flavor and their UB CC

INTERVENTIONS:
Other: very low nicotine content cigarettes — Investigational combusted cigarettes with very low nicotine content
  Other Names: VLNC
  Arms: Study EC + VLNC CC
Other: normal nicotine content cigarettes — Investigational combusted cigarettes with normal nicotine content
  Other Names: NNC
  Arms: Study EC + NNC CC
Other: Study e-cigarette — E-cigarette provided by study
  Arms: Study EC + NNC CC; Study EC + UB CC; Study EC + VLNC CC

SUMMARY:
The purpose of the study is to evaluate how limiting the nicotine content in regular cigarettes affects choices for regular cigarette and e-cigarette products. Eligible participants will be of legal age to purchase tobacco products and regularly use both e-cigarettes and regular cigarettes.

DETAILED DESCRIPTION:
Participants in this study will undergo an in-person screening session where the study will be explained in detail and participants will answer questions and provide a breath sample. During the screening session, participants will also be asked to complete surveys. Eligible participants will then complete the training procedures during which they will select an e-cigarette device to use for future preference sessions. During the 4 preference sessions, participants will sample puffs from an e-cigarette and regular cigarette and answer questions about their experience with each. They will also complete a task during which they can choose to earn puffs from the e-cigarette or regular cigarette, or choose to not take any puffs. The 4 sessions will be the same except that a different combination of e-cigarette and regular cigarette is used at each session.

ELIGIBILITY:
Inclusion Criteria:

1. Legal age to purchase tobacco products;
2. Regular user of EC and CC;
3. Owns the e-cigarette device used most often;
4. Agrees to abstain from using all tobacco products for 12 hours prior to each experimental session;
5. Self-reporting tobacco flavored e-liquid is preferred or usual flavor e-liquid

Exclusion Criteria:

1. Unstable medical conditions as determined by the licensed medical professional;
2. Unstable psychiatric conditions as determined by the licensed medical professional or PI;
3. Currently pregnant, breastfeeding, trying to become pregnant or unwilling to agree to use adequate protection to avoid pregnancy;
4. Serious quit attempt of either or both products in the past 3 months resulting in >30 days of abstinence;
5. Currently using nicotine replacement therapy or other pharmacotherapies as cessation aide;
6. Plans to quit use of either EC or CC, or all tobacco products in the next 45 days;
7. Self-reporting nicotine-free, CBD, or THC liquid is preferred or usual e-liquid;
8. Vital signs outside of the following range (participants failing for vital signs will be allowed to re-screen once):

   1. Systolic blood pressure (BP) greater than or equal to 160 mm/hg
   2. Diastolic BP greater than or equal to 100 mm/hg
   3. Heart rate greater than or equal to 115 bpm;
9. Allergy to propylene glycol or vegetable glycerin;
10. Previous adverse reaction when using vaping device or e-liquid;
11. Current or recent alcohol or drug abuse problems;
12. Previous use of SPECTRUM or other reduced nicotine content cigarettes in past 3 months;
13. Literate and able to independently complete and comprehend the consent form and other written study materials and measures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Number of choices for CC during preference task | during preference session, approximately 2 hours
  Participants will complete a preference task during which they will choose to take puffs from the session EC, the session CC, or to abstain from taking any puffs. A total of 10 trials will be completed. The number of choices for CC will be compared across the preference sessions.

SECONDARY OUTCOMES:
Number of choices for EC during preference task | during preference session, approximately 2 hours
  Participants will complete a preference task. The number of choices for EC will be compared across the preference sessions.
Number of choices to abstain during preference task | during preference session, approximately 2 hours
  Participants will complete a preference task. The number of choices to abstain from any puffs will be compared across the preference sessions.
Cigarette Evaluation Scale | during preference session, approximately 2 hours
  subjective reactions (e.g., satisfaction, dizziness) to CC product as well as how much a measure of how much they would pay for a day's worth of the product. Scale is administered on a 0-100 scale where 0 is "not at all" and 100 is "extremely"
Perceived health risk | during preference session, approximately 2 hours
  Participants will rate on a scale from 1 (very low risk) to 7 (very high risk) their perceived risk of developing a variety of health conditions (e.g., lung cancer, heart disease, stroke) as a result of using each product.
Craving | during preference session, approximately 2 hours
  craving rating on a scale from 1-10 [no urge to extremely strong urge] for CC and EC after product exposure relative to baseline value
Product Valuation | during preference session, approximately 2 hours
  Participants will be asked how many days per month would they use the CC product they just sampled at a variety of price increments
CO boost | during preference session, approximately 2 hours
  Breath carbon monoxide (CO) value after product exposure during the preference task relative to baseline value
Cross Price Elasticity | during preference session, approximately 2 hours
  the change in demand for the session CC in response to a change in price of the session EC

CONTACTS AND LOCATIONS:
Overall Officials: Francis McClernon, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No